CLINICAL TRIAL: NCT06455930
Title: Biomechanical Changes Underpinning Stand-on Ride-on Power Mobility Devices for Children With Cerebral Palsy
Brief Title: Stand-on Ride-on Power Mobility Devices for Children With Cerebral Palsy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of North Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Guilherme Cesar, Assistant Professor, University of North Florida
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNFlorida
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Power Mobility Device; Balance; Muscle activity; Mobility
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: In this foundational study, only one group will participate and receive the intervention.
Masking Description: In this phase of the study, masking cannot be done as all participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Stand-on ride-on power mobility device — Children will receive the adapted toy car (individually-adapted stand-on PMD) to take home and use for three months. PMD will be used at their house and familiar environments to the family (e.g., neighborhood, parks, schools).

SUMMARY:
The goal of this interventional study is to learn about the biomechanical factors underlying the beneficial changes in children with cerebral palsy after using individually-adapted stand-on ride-on power mobility devices (PMD).

The main questions we aim to answer are:

* How does the use of stand-on PMDs affect static balance in children with cerebral palsy?
* How does the use of stand-on PMDs affect dynamic balance and mobility function in children with cerebral palsy?

Children ages 4-6 years old with cerebral palsy (GMFCS levels II and III) will:

* Use individually-adapted stand-on PMDs for three months.
* Undergo tests to measure static balance, dynamic balance, and mobility function before and after the intervention.
* Receive a full biomechanical assessment (kinematics, kinetics, muscle activity, gait spatiotemporal characteristics).

Researchers will compare pre-intervention and post-intervention measurements to quantify improvements in balance, muscle activation, and mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spastic diplegia CP, GMFCS level III;
2. Between 4 and 6 years old (age band selected based on the benefits of early intervention and the age-limitation imposed from the size constraints of the PMDs (toy cars) selected for the intervention);
3. Able to stand and to walk short distances (at least 10 meters) with or without external assistance;
4. Physician medical clearance to participate; and
5. Exhibit sufficient cooperation and attention so that simple verbal instructions can be followed.

Exclusion Criteria:

1. Have notable orthopedic conditions (e.g., lower extremity amputation; recent hip surgeries or soft tissue lengthening);
2. Inadequate vision to complete study's procedures safely;
3. Serious/unstable cardiac conditions that prevent engagement in the Evaluation Sessions; and
4. Any other factor that might hinder full participation in the study or confound interpretation of the results.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Center of pressure sway area, standing | Baseline, Pre (3 months post Baseline), Post (3 months post Pre)
  Measure of balance control during independent standing

SECONDARY OUTCOMES:
Thigh muscle co-contraction (quadriceps:biceps femoris) | Baseline, Pre (3 months post Baseline), Post (3 months post Pre)
  Agonist-antagonist muscle efficiency during functional tasks (e.g., sit-to-stand, independent static standing).
Center of pressure sway area, sit-to-stand | Baseline, Pre (3 months post Baseline), Post (3 months post Pre)
  Measure of dynamic balance control during sit-to-stand
Trunk-pelvis coupling | Baseline, Pre (3 months post Baseline), Post (3 months post Pre)
  Quantification of timing and magnitude of whole-body motor control coordination during functional tasks (e.g., sit-to-stand, walking turns).

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Further discussion is needed given vulnerable population.